CLINICAL TRIAL: NCT05776407
Title: A Single Dose-escalation and Dose-expansion Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Allogeneic CAR-T Targeting CD19 in Patients With Refractory or Relapsed B Cell Lymphoma.
Brief Title: Safety, Efficacy and Pharmacokinetics of ThisCART19A in Patients With Refractory or Relapsed B Cell Lymphoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Collaborators: Fundamenta Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FT400-006-2
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Refractory or Relapsed B Cell Lymphoma
Keywords: Allogeneic CAR T，B cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART19A cells infusion (Experimental): In this study, allogeneic anti-CD19 CAR T cells (ThisCART19A) infusion is used to treat patients with r/r B cell Lymphoma.
  Interventions: Drug: ThisCART19A; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Drug: ThisCART19A — Single dose of Allogeneic Anti-CD19 CAR T cells (ThisCART19A) will be infused after the lymphodepletion conditioning of Fludarabine, Cyclophosphamide and Etoposide.
  Other Names: Allogeneic Anti-CD19 CAR T cells
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.
Drug: Etoposide — Etoposide is used for lymphodepletion.
  Other Names: VP-16

SUMMARY:
This is a phase 1/2, open-label study to assess the efficacy, safety and pharmacokinetics of ThisCART19A (Allogeneic Anti CD19 CAR-T) in patients with refractory or relapsed CD19 positive B cell Lymphoma.

DETAILED DESCRIPTION:
This is a phase 1/2, single-center, nonrandomized, open-label, dose-escalation and dose-expansion study to evaluate the efficacy, safety and pharmacokinetics of ThisCART19A in patients with r/r CD19 positive B cell Lymphoma and identify a treatment regimen most likely to result in clinical efficacy while maintaining a favorable safety profile. AIDS-related B-cell lymphoma were not excluded from this clinical trial.

Before initiating ThisCART19A infusion, subjects will be administered lymphodepletion chemotherapy composed of fludarabine、cyclophosphamide and VP-16. At Day 0 of the Treatment Period, subjects will receive an intravenous (IV) infusion of ThisCART19A. All subjects are monitored during the treatment period through Day 42. All subjects who receive a dose of ThisCART19A will be followed up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years ≤ age ≤ 65 years.
2. Voluntarily sign a documented IRB-approved ICF prior to any screening procedure.
3. Patients with histologically confirmed B-cell NHL defined by the World Health Organization (WHO) 2016, including but not limited to diffuse large B-cell lymphoma (DLBCL), follicular lymphoma transferring to DLBCL, mantle cell lymphoma (MCL), follicular lymphoma 3B (FL-3B), original Mediastinal (thymus) large B-cell lymphoma, high-grade B-cell lymphoma and AIDS-associated B-cell lymphoma.
4. Prior therapy must have included: Anti-CD20 monoclonal antibody and Anthracycline containing chemotherapy regimen.
5. Had available evaluation lesion.
6. ECOG(Eastern Cooperative Oncology Group) ≤ 2 or Karnofsky ≥ 60%.
7. Serum creatinine≤1.5×ULN or creatinine clearance>30 mL/min/1.73 m2.
8. Alanine aminotransferase(ALT)≤5×ULN(Upper limit of normal) and total bilirubin(TBIL)<2.0 mg/dL(for patients with Gilbert heald diseases, live involvement and taking atazanavir or indinavir, TBIL<3.0 mg/dL can be enrolled.)
9. Left ventricular ejection fraction(LVEF)≥40%
10. Absolute neutrophile counts≥1000/mm3
11. Thrombocyte≥30000/mm3
12. Total bilirubin(TBIL) ≤ 2.0 mg/dL
13. Confirmed Cluster of differentiation(CD)19 positive by biopsy for the patients who received CD19 target therapy before.
14. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
15. AIDS Related B Cell Lymphoma :HIV virus loading < 200 copy/ml and CD4+T cell counts >200 cells/mm3 within 4 weeks before screening.
16. Patients with TBIL≤ 1.5 mg/dL, Aspartate aminotransferase(AST) and ALT ≤ 3×ULN, and hepatitis B virus(HBV) DNA <2000 IU/ml can be enrolled for HBV positive patients(defined as hepatitis B virus surface antigen(HBsAg) positive and hepatitis B core(HBc)-total positive ) and hepatitis C virus(HCV) positive patients(defined as HCV antibody positive) . Patients with cirrhosis are excluded.
17. Hepatitis B core antibody(HBcAb) positive patients enrolled in this trial have to taking anti-HBV drugs during the whole research.

Exclusion Criteria:

1. Known for allergic to the preconditioning measures.
2. Uncontrollable bacterial, fungal, viral infection before enrollment.
3. Patients with pulmonary embolism within 3 months prior enrollment.
4. Intolerable serious cardiovascular and cerebrovascular diseases and hereditary diseases.
5. Imaging confirmed the presence of central nervous system involvement(including primary and secondary) and rapid progressing diseases.
6. Receive allogeneic hematopoietic stem cell transplantation less than 100 days.
7. Systemic steroid use (e.g., prednisone ≥20mg) within 3 days prior to screening. iIntermittent use of topical, inhaled or intranasal steroids recently or currently. Or systemic disease requiring long-term use of immunosuppression drugs.
8. Excluded the patients received Influenza vaccinations within 2 weeks prior to lymphodepletion (Received Severe Acute Respiratory Syndrome-Corona virus disease(SARS-COV)19 vaccines could be included. Received inactivated, live/non-live adjuvant vaccines could be enrolled).
9. Excluded women who are in pregnant or lactating, and female subjects or partners who plan to be pregnant within 1 year after infusion. Male subjects planning pregnancy within 1 year after infusion should be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) observation in patient with r/r B cell Lymphoma | 28 days
  DLT was defined as CAR T cells-related events with onset within first 28 days following infusion.
The incidence of all grade TEAEs and ≥3 grade TEAEs | Up to 2 years after ThisCART19A infusion
  Incidence of treatment-emergent adverse events (TEAEs) and ≥3 grade TEAEs
Objective Response Rate | Up to 2 years after ThisCART19A infusion
  the incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as best response to treatment.
Duration of response (DOR) | Up to 2 years after ThisCART19A infusion
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators and based on the Lugano 2014 assessment criterion for r/r B cell Lymphoma, or death regardless of cause.
Progress-free survival (PFS) | Up to 2 years after ThisCART19A infusion
  PFS is defined as the time from the ThisCART19A infusion date to the date of disease progression assessed by investigators and based on the Lugano 2014 assessment criterion, or death any cause.

SECONDARY OUTCOMES:
TTR (Time to response) | Up to 2 years after ThisCART19A infusion
  TTR is defined as the time from ThisCART19A infusion to first assessed CR or PR based on the Lugano 2014 assessment criterion.
OS (Overall survival) | Up to 2 years after lymphodepletion
  Overall survival (OS) is defined as the time from the date of lymphodepletion until death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No